CLINICAL TRIAL: NCT03145909
Title: A Phase 1 Study Evaluating the Safety, Pharmacokinetics and Anti-Tumor Activity of ABBV-176 in Subjects With Advanced Solid Tumors Likely to Express Prolactin Receptor (PRLR)
Brief Title: A Study Evaluating the Safety, Pharmacokinetics and Anti-Tumor Activity of ABBV-176 in Subjects With Advanced Solid Tumors Likely to Express Prolactin Receptor (PRLR)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Safety
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M15-916; 2016-004597-18 (EudraCT Number)
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Advanced Solid Tumors Cancer
Keywords: Cancer; Metastatic; Prolactin Receptor (PRLR); Breast cancer; Colorectal cancer; Adrenocortical carcinoma,; Chromophobe renal cell carcinoma; Hepatocellular carcinoma
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Breast Neoplasms; Colorectal Neoplasms; Adrenocortical Carcinoma; Carcinoma, Renal Cell; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation Cohort (Experimental): ABBV-176 will be administered via intravenous infusion at escalating dose levels until the maximum tolerated dose is reached.
  Interventions: Drug: ABBV-176
- Expanded RPTD Cohort (Experimental): ABBV-176 via intravenous administration in participants with breast cancer at the Recommended Phase Two Dose (RPTD) determined during the Dose Escalation Cohort
  Interventions: Drug: ABBV-176

INTERVENTIONS:
Drug: ABBV-176 — Intravenous infusion

SUMMARY:
This is an open-label, Phase I, dose-escalation study to determine the maximum tolerated dose (MTD) and the recommended phase two dose (RPTD), and to assess the safety, preliminary efficacy, and pharmacokinetic (PK) profile of ABBV-176 for participants with advanced solid tumors likely to express Prolactin Receptor (PRLR). The study will consist of 2 cohorts: Dose Escalation and Expanded Recommended Phase 2 Dose.

ELIGIBILITY:
Inclusion Criteria:

* Participant has histological confirmation of a locally advanced or metastatic solid tumor of a type associated with Prolactin Receptor (PRLR) expression that has progressed on prior treatment, is not amenable to treatment with curative intent, and has no other therapy options known to provide clinical benefit or the subject is ineligible for such therapies.
* Dose Escalation Cohort: must have breast cancer, colorectal cancer, adrenocortical carcinoma, chromophobe renal cell carcinoma.
* Expanded Cohort: must have breast cancer.
* Participant must consent to provide the following for biomarker analyses:
* Dose Escalation Cohort: archived tumor tissue or fresh tumor biopsy.
* Expanded Cohort: archived tumor tissue and fresh tumor biopsy.
* Participant has Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Participant has adequate bone marrow, renal, and hepatic function.

Exclusion Criteria:

* Participant received anticancer therapy including chemotherapy, immunotherapy, radiotherapy, biologic, or any investigational therapy within 21 days before Study Day 1; participant received palliative radiotherapy or small molecule targeted anti-cancer agents within 14 days of Study Day 1.
* Participant has prior exposure to any pyrrolobenzodiazopine-containing agent
* Participant has unresolved, clinically significant toxicities from prior anticancer therapy, defined as greater than Grade 1 on Common Terminology for adverse events.
* Participant has clinically significant uncontrolled conditions.
* Participant has a history of major immunologic reaction to any Immunoglobulin G (IgG).
* Participant has received more than 4 prior lines of systemic cytotoxic therapy (not including neo-adjuvant or adjuvant therapy).

  * For prior cytotoxic therapy, treatment for 1 full cycle or less will not be considered as prior therapy unless the patient experienced progression of disease while on that therapy.
* Participant has a history of >= grade 3 AST, ALT, or bilirubin increase or has extensive liver resection (i.e., left lobe resection).
* Participant has a history of cholecystitis (subject with history of cholecystectomy will not be excluded), or has active gallbladder disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Dose Escalation Cohort: Tmax of ABBV-176 | Up to approximately 57 days
  Time to Cmax (Tmax) of ABBV-176
Dose Escalation Cohort: AUC∞ for ABBV-176 | Up to approximately 57 days
  AUC∞ is the area under the plasma concentration-time curve from Time 0 to infinite time.
Dose Escalation Cohort: Terminal phase elimination rate constant (β) for ABBV-176 | Up to approximately 57 days
  Terminal phase elimination rate constant (β)
Dose Escalation Cohort: Recommended Phase 2 dose (RPTD) for ABBV-176 | Minimum first cycle of dosing (up to 21 days)
  The RPTD will be determined using available safety and pharmacokinetics data upon completion of the Dose Escalation Cohort.
Dose Escalation Cohort: Cmax of ABBV-176 | Up to approximately 57 days
  Maximum observed plasma concentration (Cmax) of ABBV-176.
Dose Escalation Cohort: Maximum tolerated dose (MTD) of ABBV-176 | Minimum first cycle of dosing (up to 21 days)
  MTD will be defined as the highest dose level at which less than or equal to 33% of participants experience a dose limiting toxicity.
Expanded Recommended Phase Two Dose (RPTD) Cohort: Objective Response Rate (ORR) | Up to approximately 2 years
  ORR is defined as the proportion of participants with a response of partial response (PR) or better per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
Dose Escalation Cohort: AUCt for ABBV-176 | Up to approximately 57 days
  Area Under the Plasma Concentration-time Curve from Time 0 to the Time of the Last Measurable Concentration (AUCt) for ABBV-176.
Dose Escalation Cohort: t1/2 for ABBV-176 | Up to approximately 57 days
  Terminal elimination half-life (t1/2)

SECONDARY OUTCOMES:
Expanded RPTD Cohort: AUCt for ABBV-176 | Up to approximately 15 days
  Area Under the Plasma Concentration-time Curve from Time 0 to the Time of the Last Measurable Concentration (AUCt)
Expanded RPTD Cohort: Tmax of ABBV-176 | Up to approximately 15 days
  Time to Cmax (Tmax) of ABBV-176
Expanded RPTD Cohort: Overall Survival (OS) | Up to 2 years after the last dose of study drug
  OS is defined as number of days from the date of the first dose to the date of death for all dosed subjects. For subjects who are not deceased, the data will be censored at the date of the last study visit, or the last know date to be alive, whichever is later.
Expanded RPTD Cohort: Cmax of ABBV-176 | Up to approximately 15 days
  Maximum observed plasma concentration (Cmax) of ABBV-176.
Expanded RPTD Cohort: Duration of Response (DOR) | Up to approximately 2 years
  DOR is defined as the time from the date of the participant's documented first response of PR or better to the date of documented disease progression or death due to the disease, whichever occurs first.
Expanded RPTD Cohort: Terminal phase elimination rate constant (β) for ABBV-176 | Up to approximately 15 days
  Terminal phase elimination rate constant (β) for ABBV-176
Expanded Recommended Phase Two Dose (RPTD) Cohort: Progression-Free Survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the participant's first dose of study drug (Day 1) to the date of documented disease progression (per RECIST 1.1), or death due to any cause, whichever occurs first.
Expanded RPTD Cohort: Change in ECOG Performance Status | Up to approximately 2 years
  Change from baseline in Eastern Cooperative Oncology Group (ECOG) Performance Status
Expanded RPTD Cohort: AUC∞ for ABBV-176 | Up to approximately 15 days
  Area Under the Plasma Concentration-time Curve from Time 0 to infinite time (AUC∞)
Expanded RPTD Cohort: t1/2 for ABBV-176 | Up to approximately 15 days
  Terminal elimination half-life (t1/2) for ABBV-176
Dose Escalation Cohort: Change from Baseline in QTcF | Up to approximately 47 days
  QT interval measurement corrected by Fridericia's formula (QTcF) mean change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (11):
- United States (7):
  - HonorHealth Research Institute - Pima /ID# 161078, Scottsdale, Arizona
  - City of Hope /ID# 161079, Duarte, California
  - Yale University /ID# 201357, New Haven, Connecticut
  - St. Lukes Cancer Institute /ID# 201353, Kansas City, Missouri
  - Washington University-School of Medicine /ID# 162745, St Louis, Missouri
  - Rutgers Cancer Institute of NJ /ID# 161080, New Brunswick, New Jersey
  - University of Utah /ID# 161606, Salt Lake City, Utah
- Australia (2):
  - Sydney Children's Hospital /ID# 162917, Randwick, New South Wales
  - Mater Misericordiae /ID# 162918, South Brisbane, Queensland
- Rigshospitalet /ID# 159707, Copenhagen Ø, Capital Region, Denmark
- Hosp Univ Madrid Sanchinarro /ID# 161644, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lemech C, Woodward N, Chan N, Mortimer J, Naumovski L, Nuthalapati S, Tong B, Jiang F, Ansell P, Ratajczak CK, Sachdev J. A first-in-human, phase 1, dose-escalation study of ABBV-176, an antibody-drug conjugate targeting the prolactin receptor, in patients with advanced solid tumors. Invest New Drugs. 2020 Dec;38(6):1815-1825. doi: 10.1007/s10637-020-00960-z. Epub 2020 Jun 10. PMID 32524319